CLINICAL TRIAL: NCT05024292
Title: Oriental Research Alliance of Acute Ischemic Stroke Given Endovascular Treatment: Technique Feasibility, Safety and Neuroprotective Effects of in Situ Ischemic Postconditioning in Patients Underwent Successful Endovascular Thrombectomy
Brief Title: Oriental Research AlliaNce of Acute Ischemic Stroke Given Endovascular Treatment
Acronym: ORANGE
Status: Recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Collaborators: Zhangzhou Municipal Hospital of Fujian Province (Other)
Responsible Party: Principal Investigator, Yueqi Zhu, Associated dean of the radiology, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Other Study IDs: 2021MT
Record Dates: First submitted 2021-08-22; First posted 2021-08-27 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Ischemic Stroke
Keywords: acute ischemic stroke; thrombectomy; thrombolysis; outcome
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — thrombus retrieved from the occluded artery. Serum collected from the vein at different time points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- rapid local ischemic postconditioning (RL-IPostC) group: RL-IPostC is performed immediately after successful reperfusion with 5 circules of balloon inflations in the ipsilateral internal carotid artery, each circulation includes inflation lasting 15 seconds followed by 15 seconds of deflation.
  Interventions: Procedure: rapid local ischemic postconditioning (RL-IPostC)
- control group: no intervention was provided after successful reperfusion

INTERVENTIONS:
Procedure: rapid local ischemic postconditioning (RL-IPostC) — with 5 circules of balloon inflations in the ipsilateral internal carotid artery, each circulation includes inflation lasting 15 seconds followed by 15 seconds of deflation
  Groups: rapid local ischemic postconditioning (RL-IPostC) group

SUMMARY:
To determine the safety and efficacy of in situ ischemic postconditioning immediately after successful reperfusion in AIS patients underwnet EVT.

DETAILED DESCRIPTION:
For acute ischemic stroke (AIS) patients with large vessel occlusion in the anterior circulation receieved successful reperfusion, in situ ischemic postconditioning (ISIPC) was performed immediately after successful reperfusion with 5 circules of balloon inflations in the ipsilateral internal carotid artery, each circulation includes inflation lasting 15 seconds followed by 15 seconds of deflation.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age ≥ 18 to 95 years) patients with an occlusion of the internal carotid artery or M1 or M2 segment of the middle cerebral artery,;
2. Patients with a score of at least 6 on the National Institutes of Health Stroke Scale (NIHSS) at admission and a score of 0 or 1 on the modified Rankin scale before the onset of stroke;
3. Patients with a score of at least 6 on the Alberta Stroke Program Early CT score (ASPECTS) value;
4. Baseline multimodal-CT imaging, including NCCT, CTA and CTP, performed at the trial-site hospital
5. The modified thrombolysis in cerebral infarction (mTICI) scale 2b to 3 achieved in the infarct-related artery after the last thrombectomy attempt

Exclusion Criteria:

1. Stoke of large artery atherosclerotic origin or other determined factors (such as dissection) or tandem occlusion;
2. Patients underwent rescue angioplasty or stenting after thrombectomy

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were treated according to national guidelines for treatment of AIS, including intravenous thrombolysis, if indicated. Thrombectomy were performed according to standard techniques. The method of endovascular therapy was selected at the discretion of treating physicians and could include stent retriever and/or catheter aspiration.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
functional independence | 3 month
  mRS 0-2

SECONDARY OUTCOMES:
excellent functional independence | 3 month
  mRS 0-1
early therapeutic response | on day 5, 6, or 7 of hospitalization or at discharge if it occurred before day 5
  defined as a decrease in the NIHSS score of ≥10 from baseline or an NIHSS score of 0 or 1
Mortality | 3 month
  Mortality of 3 month after stoke onset
hemorrhagic transformation | 24 hours after treatment
  according to European Cooperative Acute Stroke Study II criteria
Symptomatic intracerebral hemorrhage (sICH) | 24 hours after treatment
  an increase of ≥4 points on the National Institutes of Health Stroke Scale (NIHSS) according to Heidelberg Bleeding Classification
malignant infarction | 24 hours after treatment
  defined as infarct lesions with significant space-occupying mass effect with over 1/2 affected middle cerebral artery territory with imaging signs of herniation and/or and clinical signs of herniation requiring decompressive hemicraniectomy and/or leading to death due to direct implications of stroke

CONTACTS AND LOCATIONS:
Overall Officials: Yueqi Zhu, PhD, Study Chair — Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Locations (2):
- China (2):
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou, Fujian
  - Shanghai Sixth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided